CLINICAL TRIAL: NCT03884062
Title: Clinical Impacts of Achieving Sustained Virological Response in Patients With Advanced Hepatic Fibrosis Related to Chronic HCV Treated With Direct Acting Antivirals
Brief Title: Clinical Impacts of Achieving SVR in Patients With Advanced Hepatic Fibrosis Related to Chronic HCV Treated With Direct Acting Antivirals
Status: Completed | Type: Observational
Sponsor: Egyptian Liver Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HCV-DAA
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: HCC in Chronic HCV Patients With Advanced Liver Fibrosis
Keywords: HCC, chronic hepatitis C, hepatitis C, liver fibrosis
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DAAs-SVR.: annual incidence of HCC in chronic hepatitis C patients with advanced liver fibrosis (F3 and F4) after achieving DAAs-SVR.
  Interventions: Drug: DAAs

INTERVENTIONS:
Drug: DAAs — lab, U/S, Fibroscan & CT if needed

SUMMARY:
Chronic HCV infection has relatively slow rate of progression. Liver fibrosis is the main sequlae and usually progressed to cirrhosis after long period (10 to 20 years) [6]. Once cirrhosis is established the disease progression remains unpredictable: cirrhosis can remain indolent for many years in some patients whilst progressing in others to HCC, hepatic decompensation and death. Overall once cirrhosis has developed there is a 1-5% annual risk of HCC and a 3-6% annual risk of hepatic decompensation. Following an episode of decompensation the risk of death in the following year is between 15% and 20% Treatment of chronic HCV has been dramatically changed in the last few years with introduction of direct acting antivirals (DAAs). The new therapies with excellent safety profiles, shorter duration of therapy and marked higher efficacy can be even used in patients with advanced fibrosis and cirrhosis

DETAILED DESCRIPTION:
Chronic HCV infection has relatively slow rate of progression. Liver fibrosis is the main sequlae and usually progressed to cirrhosis after long period (10 to 20 years) [6]. Once cirrhosis is established the disease progression remains unpredictable: cirrhosis can remain indolent for many years in some patients whilst progressing in others to HCC, hepatic decompensation and death. Overall once cirrhosis has developed there is a 1-5% annual risk of HCC and a 3-6% annual risk of hepatic decompensation. Following an episode of decompensation the risk of death in the following year is between 15% and 20% Treatment of chronic HCV has been dramatically changed in the last few years with introduction of direct acting antivirals (DAAs). The new therapies with excellent safety profiles, shorter duration of therapy and marked higher efficacy can be even used in patients with advanced fibrosis and cirrhosis

ELIGIBILITY:
Inclusion Criteria:

* above 12 years old
* fibroscan F3 or F4
* HCV positive
* Received DAAs

Exclusion Criteria:

* below 12 years old
* fibroscan below F3
* HCV negative

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all subjects from screening with positive HCV whom received treatment for 12/24 week with DAAs
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Detection of HCC by CT | 12-45 months after SVR
  incidence of HCC in chronic hepatitis C patients with advanced liver fibrosis (F3 and F4) after achieving DAAs-SVR

SECONDARY OUTCOMES:
fibrosis stage changes by Fibroscan | 12-45 months after SVR
  post treatment fibrosis stage in chronic hepatitis C patients with advanced liver fibrosis (F3 and F4) after achieving DAAs-SVR

IPD SHARING:
Plan to Share IPD: No